CLINICAL TRIAL: NCT00406315
Title: A Sixteen-Week, Multi-Center, Open-Label Study Evaluating The Safety, Tolerability, And Efficacy Of Switching From Quetiapine To Ziprasidone In Subjects Diagnosed With Schizophrenia Or Schizoaffective Disorder
Brief Title: Study Evaluating The Safety, Tolerability, And Efficacy Of Switching From Quetiapine To Ziprasidone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281148
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: ziprasidone, quetiapine (Seroquel) switch, open label, flexible dose, schizophrenia, schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A1 (Other): atypical antipsychotic for the treatment of schizophrenia
  Interventions: Drug: ziprasidone

INTERVENTIONS:
Drug: ziprasidone — Days 1-3: 40 mg twice a day (BID); Days 4-7: 60 mg BID; Day 8: 80 mg BID; Flexible dose between 40-80 mg BID (adjustable up to 40 mg daily/week) for the remainder of the 16-week treatment phase and continuing throughout the 16-week follow-up phase
  Other Names: Geodon, Zeldox

SUMMARY:
The primary objective of this study is to evaluate change in weight as a result of switching from quetiapine to ziprasidone, in subjects with schizophrenia or schizoaffective disorder who have failed to achieve a satisfactory clinical response to quetiapine due to lack of efficacy or poor tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, between 18 and 55 years of age, at the time of consent.
* Subjects must have a primary diagnosis of schizophrenia, any subtype (code 295.xx), or schizoaffective disorder as defined in DSM-IV-TR (Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition)
* Subjects must have normal vital signs, physical examination, ECG, and laboratory findings except for minor deviations determined and documented to be clinically insignificant by the investigator or a sub-investigator who is a medical doctor.

Exclusion Criteria:

* Subjects who are unable to provide informed consent
* Subjects who meet criteria for a DSM-IV-TR Axis I (Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition) diagnosis other than schizophrenia or schizoaffective disorder, including psychoactive substance abuse or dependence within one year of study entry
* Females who are pregnant, breast feeding, or lactating at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (26):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Costa Mesa, California
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Temecula, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Hialeah, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Des Plaines, Illinois
  - Pfizer Investigational Site, Oakbrook Terrace, Illinois
  - Pfizer Investigational Site, Schaumburg, Illinois
  - Pfizer Investigational Site, Topeka, Kansas
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Nashua, New Hampshire
  - Pfizer Investigational Site, Olean, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Bothell, Washington
  - Pfizer Investigational Site, Kirkland, Washington
- Brazil (3):
  - Pfizer Investigational Site, Aparecida de Goiânia, Goiás
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, São Paulo, São Paulo
- Germany (4):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Düsseldorf
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, München
- Greece (2):
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Thessaloniki
- Pfizer Investigational Site, Zamora, Spain
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, İzmit

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281148&StudyName=Study%20Evaluating%20The%20Safety%2C%20Tolerability%2C%20And%20Efficacy%20Of%20Switching%20From%20Quetiapine%20To%20Ziprasidone

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An additional 14 subjects had a baseline visit but were never treated.
Groups:
- Ziprasidone: For Days 1 to 3, the subject was dosed at 40 mg twice a day (BID) (80 mg/day), taking two 20 mg capsules BID. For Days 4 to 7, the subject was dosed at 60 mg BID (120 mg/day), taking one 60 mg capsule BID. On Day 8, the subject was dosed at 80 mg BID (160 mg/day), taking one 20 mg capsule and one 60 mg capsule BID. Based on clinical judgment, the dose could have been adjusted once per week in increments/decrements of up to 40 mg daily.
Period: Overall Study
Arm/Group | Ziprasidone
Started | 241 (Started = Treated)
Completed | 100
Not Completed | 141
Not completed — Death | 1
Not completed — Adverse Event | 39
Not completed — Laboratory Abnormality | 4
Not completed — Lack of Efficacy | 13
Not completed — Other | 33
Not completed — Lost to Follow-up | 21
Not completed — Withdrawal by Subject | 30

BASELINE CHARACTERISTICS:
Arm/Group | Ziprasidone
Number analyzed (Participants) | 241
Age, Customized [Number; unit: participants]
  < 18 years | 0
  18 to 44 years | 140
  45 to 64 years | 101
  > = 65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 130

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight at Week 16
Description: Weight value: Change = value at Week 16 or Week 16 Last Observation Carried Forward (LOCF) minus value at Baseline.
Time Frame: Baseline, Week 16, Week 16 LOCF
Population: Safety population = all enrolled subjects who took at least 1 dose of study medication. LOCF was used to impute missing values. LOCF value was the last non-missing, post-baseline observation carried forward for each subject.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Ziprasidone
Number analyzed (Participants) | 231
kilogram
  Week 16 (n=133) | -1.09 (3.918)
  Week 16 LOCF (n=231) | -0.73 (3.725)
Statistical Analysis 1: Comparison: Ziprasidone; Week 16; Test type: Superiority or Other; One-sided upper confidence limit = -0.53 — A one-sided 95% confidence interval (CI) was constructed for the mean weight change from baseline to infer whether there was a significant decrease in weight
Statistical Analysis 2: Comparison: Ziprasidone; Week 16 LOCF. Based on past information, the standard deviation of the mean weight difference was expected to be 2.2. The sample size of the study was estimated so that the one-sided CI of the mean weight decrease has a certain width. To obtain a one-sided CI with a width of 0.27 kg, a sample size of 180 subjects was needed. In other words, we were 95% certain that the true mean weight decrease was in an interval starting from the observed weight decrease and extending 0.27 kg unit above it; Test type: Superiority or Other; One-sided upper confidence limit = -0.33 — A one-sided 95% CI was constructed for the mean weight change from baseline to infer whether there was a significant decrease in weight

2. Secondary Outcome: Change From Baseline in Fasting Lipid Profile (Total Cholesterol) at Week 16
Description: Total cholesterol value: Change = value at Week 16 minus value at Baseline.
Time Frame: Baseline, Week 16
Population: Safety population.
Measure: Mean (Standard Deviation); unit: milligram (mg)/deciliter (dL)
Arm/Group | Ziprasidone
Number analyzed (Participants) | 128
milligram (mg)/deciliter (dL) | -3.0 (31.14)
Statistical Analysis 1: Comparison: Ziprasidone; Week 16. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -3.0, 95% CI 2-sided [-8.48 to 2.41]

3. Secondary Outcome: Change From Baseline in High-Density Lipoprotein (HDL), Low-Density Lipoprotein (LDL), and Triglycerides at Week 16
Description: HDL, LDL, and triglyceride value: Change = value at Week 16 minus value at Baseline.
Time Frame: Baseline, Week 16
Population: Safety population.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ziprasidone
Number analyzed (Participants) | 128
mg/dL
  HDL (n=128) | -0.2 (9.32)
  LDL (n=123) | -2.5 (25.66)
  Triglycerides (n=128) | -1.6 (84.58)
Statistical Analysis 1: Comparison: Ziprasidone; HDL. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -0.2, 95% CI 2-sided [-1.82 to 1.44]
Statistical Analysis 2: Comparison: Ziprasidone; LDL. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -2.5, 95% CI 2-sided [-7.07 to 2.09]
Statistical Analysis 3: Comparison: Ziprasidone; Triglycerides. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -1.6, 95% CI 2-sided [-16.44 to 13.15]

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) at Week 16
Description: HbAlc value: Change = value at Week 16 minus value at Baseline.
Time Frame: Baseline, Week 16
Population: Safety population.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Ziprasidone
Number analyzed (Participants) | 127
percent | 0.1 (0.44)
Statistical Analysis 1: Comparison: Ziprasidone; The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 0.1, 95% CI 2-sided [-0.02 to 0.14]

5. Secondary Outcome: Change From Baseline in Fasting Glucose at Week 16
Description: Fasting glucose value: Change = value at Week 16 minus value at Baseline.
Time Frame: Baseline, Week 16
Population: Safety population.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ziprasidone
Number analyzed (Participants) | 128
mg/dL | 3.0 (17.84)
Statistical Analysis 1: Comparison: Ziprasidone; The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 3.0, 95% CI 2-sided [-0.09 to 6.15]

6. Secondary Outcome: Change From Baseline in Fasting Insulin at Week 16
Description: Fasting insulin value: Change = value at Week 16 minus value at Baseline.
Time Frame: Baseline, Week 16
Population: Safety population.
Measure: Mean (Standard Deviation); unit: microinternational (mciu)/milliliter(mL)
Arm/Group | Ziprasidone
Number analyzed (Participants) | 118
microinternational (mciu)/milliliter(mL) | 134.8 (851.28)
Statistical Analysis 1: Comparison: Ziprasidone; The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 134.8, 95% CI 2-sided [-20.43 to 289.98]

7. Secondary Outcome: Change From Baseline in Waist and Hip Circumference at Week 16
Description: Waist and hip circumference value: Change = value at Week 16 minus value at Baseline.
Time Frame: Baseline, Week 16
Population: Safety population.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Ziprasidone
Number analyzed (Participants) | 132
centimeter
  Waist (n=132) | -2.9 (17.53)
  Hip (n=131) | -3.0 (18.21)
Statistical Analysis 1: Comparison: Ziprasidone; Waist. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -2.9, 95% CI 2-sided [-5.93 to 0.11]
Statistical Analysis 2: Comparison: Ziprasidone; Hip. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -3.0, 95% CI 2-sided [-6.20 to 0.10]

8. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score, Global Severity Score, and Global Incapacitation Score at Week 16
Description: AIMS: a 12-item clinician administered instrument assessing observed abnormal movements in different parts of body. Ten items scored on a 5-point scale (0 = none/normal, 4 = severe) evaluate abnormal movements in three main anatomic areas (orofacial area, extremities, and trunk). Two items are yes/no questions regarding dentures. Total scores range from 0 to 42. Item 8 indicates severity, item 9 indicates Incapacitation. AIMS total, global severity, or global incapacitation score: Change = score at Week 16 minus score at Baseline.
Time Frame: Baseline, Week 16
Population: Safety population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 144
scores on a scale
  AIMS Total Score | 0.05 (2.251)
  AIMS Global Severity Score | 0.03 (0.472)
  AIMS Global Incapacitation Score | 0.01 (0.383)
Statistical Analysis 1: Comparison: Ziprasidone; Total Score. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 0.05, 95% CI 2-sided [-0.32 to 0.42]
Statistical Analysis 2: Comparison: Ziprasidone; Global Severity Score. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 0.03, 95% CI 2-sided [-0.05 to 0.11]
Statistical Analysis 3: Comparison: Ziprasidone; Global Incapacitation Score. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 0.01, 95% CI 2-sided [-0.06 to 0.07]

9. Secondary Outcome: Change From Baseline in Positive and Negative Symptoms of Schizophrenia (PANSS) Total Score, and Positive and Negative Subscale Scores at Week 16
Description: PANSS measures severity of psychopathology in subjects with schizophrenia, schizoaffective disorder and other psychotic disorders. It includes 3 scales and a total of 30 items: 7 items comprise the positive scale, 7 comprise the negative scale, and 16 items measure general psychopathology. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210. PANSS total score and positive and negative scores: Change = score at Week 16 or Week 16 LOCF minus score at Baseline.
Time Frame: Baseline, Week 16, Week 16 LOCF
Population: Intent-to-treat population (ITT) = all enrolled subjects with baseline and at least 1 post baseline efficacy evaluation. LOCF was used to impute missing values. LOCF value was the last non-missing, post-baseline observation carried forward for each subject.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 231
scores on a scale
  Total Score, Week 16 (n=144) | -10.22 (15.027)
  Total Score, Week 16 LOCF (n=231) | -6.61 (15.306)
  Positive Subscale Score, Week 16 (n=144) | -3.30 (4.658)
  Positive Subscale Score, Week 16 LOCF (n=231) | -2.43 (4.634)
  Negative Subscale Score, Week 16 (n=144) | -1.67 (4.147)
  Negative Subscale Score, Week 16 LOCF (n=231) | -0.92 (4.373)
Statistical Analysis 1: Comparison: Ziprasidone; Total Score, Week 16. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -10.22, 95% CI 2-sided [-12.70 to -7.75]
Statistical Analysis 2: Comparison: Ziprasidone; Total Score, Week 16 LOCF. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -6.61, 95% CI 2-sided [-8.59 to -4.63]
Statistical Analysis 3: Comparison: Ziprasidone; Positive Subscale Score, Week 16. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -3.30, 95% CI 2-sided [-4.07 to -2.53]
Statistical Analysis 4: Comparison: Ziprasidone; Positive Subscale Score, Week 16 LOCF. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -2.43, 95% CI 2-sided [-3.03 to -1.83]
Statistical Analysis 5: Comparison: Ziprasidone; Negative Subscale Score, Week 16. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -1.67, 95% CI 2-sided [-2.36 to -0.99]
Statistical Analysis 6: Comparison: Ziprasidone; Negative Subscale Score, Week 16 LOCF. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -0.92, 95% CI 2-sided [-1.48 to -0.35]

10. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity Scale (CGI-S) at Week 16
Description: The CGI-S is a single item, clinician-rated scale that assesses the global severity of the subject's overall illness. The CGI-S ratings range from 1 (normal, not at all ill) to 7 (among the most severely ill subjects). CGI-S score: Change: score at Week 16 or Week 16 LOCF minus score at Baseline.
Time Frame: Baseline, Week 16, Week 16 LOCF
Population: ITT. LOCF was used to impute missing values. The LOCF value was the last non-missing, post-baseline observation carried forward for each subject.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 231
scores on a scale
  Week 16 (n=135) | -0.76 (0.868)
  Week 16 LOCF (n=231) | -0.47 (0.848)
Statistical Analysis 1: Comparison: Ziprasidone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Mean = -0.76, 95% CI 2-sided [-0.90 to -0.61]
Statistical Analysis 2: Comparison: Ziprasidone; Week 16 LOCF. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -0.47, 95% CI 2-sided [-0.58 to -0.36]

11. Secondary Outcome: Observed Cases of Clinical Global Impression Improvement Scale (CGI-I) Scores at Week 16
Description: The CGI-I is a 7-point, single-item, clinician-rated scale that assesses global improvement in the subject's clinical state in response to study treatment, and as compared to their status at pre-treatment baseline. Possible CGI-I scores range from 1 (very much improved) to 4 (no change) to 7 (very much worse).
Time Frame: Week 16, Week 16 LOCF
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 231
scores on a scale
  Week 16 (n=135) | 2.7 (1.05)
  Week 16 LOCF (n=231) | 3.2 (1.22)
Statistical Analysis 1: Comparison: Ziprasidone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Mean = 2.7, 95% CI 2-sided [2.52 to 2.88]
Statistical Analysis 2: Comparison: Ziprasidone; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; Mean = 3.2, 95% CI 2-sided [3.02 to 3.34]

12. Secondary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) Total Score at Week 16
Description: The CDSS is a 9-item, clinician-rated scale validated for rating the severity of depressive symptoms in subjects diagnosed with schizophrenia, and independent of confounding negative and extrapyramidal symptoms. The CDSS rates the severity of depressive symptoms on a 4-point scale ranging from 0 (absent) to 3 (severe). The CDSS depression total score is obtained by adding each of the item scores. Total possible score ranges from 0 to 27. CDSS possible total score: Change: score at Week 16 or Week 16 LOCF minus score at Baseline.
Time Frame: Baseline, Week 16, Week 16 LOCF
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 231
scores on a scale
  Week 16 (n=144) | -2.55 (4.364)
  Week 16 LOCF (n=231) | -1.58 (4.526)
Statistical Analysis 1: Comparison: Ziprasidone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Mean = -2.55, 95% CI 2-sided [-3.27 to -1.83]
Statistical Analysis 2: Comparison: Ziprasidone; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; Mean = -1.58, 95% CI 2-sided [-2.16 to -0.99]

13. Secondary Outcome: Change From Baseline in Schizophrenia Cognition Rating Scale (SCoRS) Total Score and Global Rating at Week 16
Description: The SCoRS is a 20-question rating scale completed via interviews with the subject and an informant, focusing on cognitive impairment and its impact on daily functioning. Each question was completed using a 4-point scale (ranging from 1=none to 4=severe). Total possible score ranged from 20 to 80. At the end of the 20 questions, the interviewer completed a Global Scale of 1-10, rating subject's overall difficulty. Higher scores on both indicated greater cognitive impairment. SCoRS total score and global rating: Change: score at Week 16 or Week 16 LOCF minus score at Baseline.
Time Frame: Baseline, Week 16, Week 16 LOCF
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 169
scores on a scale
  Total Score, Week 16 (n=137) | -4.61 (7.981)
  Total Score, Week 16 LOCF (n=169) | -4.21 (8.961)
  Global Rating, Week 16 (n=137) | -1.02 (1.708)
  Global Rating, Week 16 LOCF (n=169) | -0.88 (1.643)
Statistical Analysis 1: Comparison: Ziprasidone; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; Mean = -4.61, 95% CI 2-sided [-5.95 to -3.26]
Statistical Analysis 2: Comparison: Ziprasidone; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; Mean = -4.21, 95% CI 2-sided [-5.57 to -2.85]
Statistical Analysis 3: Comparison: Ziprasidone; Global Rating, Week 16. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -1.02, 95% CI 2-sided [-1.31 to -0.73]
Statistical Analysis 4: Comparison: Ziprasidone; Global Rating, Week 16 LOCF. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = -0.88, 95% CI 2-sided [-1.13 to -0.63]

14. Secondary Outcome: Change From Baseline in Global Assessment of Function Scale (GAF) Score at Week 16
Description: GAF Scale measures the severity of illness-related impairment in psychological, social, and occupational functioning using a 100-point scale. Total possible score ranges from 0 (not enough information available to provide GAF) to 100 (Superior functioning in a wide range of activities, life's problems never seem to get out of hand, is sought out by others because of his or her many qualities. No symptoms). The assessment was done by a trained assessor. GAF scale score: Change: score at Week 16 or Week 16 LOCF minus score at Baseline.
Time Frame: Baseline, Week 16, Week 16 LOCF
Population: ITT. LOCF was used to impute missing values. LOCF value was the last non-missing, post-baseline observation carried forward for each subject.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 230
scores on a scale
  Week 16 (n=145) | 7.88 (11.029)
  Week 16 LOCF (n=230) | 5.27 (10.626)
Statistical Analysis 1: Comparison: Ziprasidone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Mean = 7.88, 95% CI 2-sided [6.07 to 9.69]
Statistical Analysis 2: Comparison: Ziprasidone; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; Mean = 5.27, 95% CI 2-sided [3.89 to 6.65]

15. Secondary Outcome: Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TQSM) Effectiveness, Side Effect, Convenience, and Global Satisfaction Subscales at Week 16
Description: The TSQM is a 13-item subject-rated scale that evaluates the effectiveness, side effects and convenience of the medication over the past 2-3 weeks. Likert scale: 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Somewhat Dissatisfied, 4=Neither Satisfied Nor Dissatisfied, 5=Somewhat Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. Worst value is 0 and best value is 100. TSQM Effectivenss, Side Effect, Convenience, and Global Satisfaction scores: Change: score at Week 16 or Week 16 LOCF minus score at Baseline.
Time Frame: Baseline, Week 16, Week 16 LOCF
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 180
scores on a scale
  Effectiveness, Week 16 (n=178) | 10.49 (30.662)
  Effectiveness, Week 16 LOCF (n=178) | 10.49 (30.662)
  Side Effect, Week 16 (n=167) | 18.49 (42.883)
  Side Effect, Week 16 LOCF (n=167) | 18.49 (42.883)
  Convenience, Week 16 (n=180) | 6.45 (23.630)
  Convenience, Week 16 LOCF (n=180) | 6.45 (23.630)
  Global Satisfaction, Week 16 (n=179) | 15.32 (36.304)
  Global Satisfaction, Week 16 LOCF (n=179) | 15.32 (36.304)
Statistical Analysis 1: Comparison: Ziprasidone; Effectiveness, Week 16. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 10.49, 95% CI 2-sided [5.95 to 15.02]
Statistical Analysis 2: Comparison: Ziprasidone; Effectiveness, Week 16 LOCF. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 10.49, 95% CI 2-sided [5.95 to 15.02]
Statistical Analysis 3: Comparison: Ziprasidone; Side Effect, Week 16. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 18.49, 95% CI 2-sided [11.94 to 25.04]
Statistical Analysis 4: Comparison: Ziprasidone; Side Effect, Week 16 LOCF. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 18.49, 95% CI 2-sided [11.94 to 25.04]
Statistical Analysis 5: Comparison: Ziprasidone; Convenience, Week 16. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 6.45, 95% CI 2-sided [2.98 to 9.93]
Statistical Analysis 6: Comparison: Ziprasidone; Convenience, Week 16 LOCF. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 6.45, 95% CI 2-sided [2.98 to 9.93]
Statistical Analysis 7: Comparison: Ziprasidone; Global Satisfaction, Week 16. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 15.32, 95% CI 2-sided [9.97 to 20.68]
Statistical Analysis 8: Comparison: Ziprasidone; Global Satisfaction, Week 16 LOCF. The arithmetic mean and the corresponding 2-sided 95% CI are reported. All CIs are unadjusted for any multiplicity; Test type: Superiority or Other; Mean = 15.32, 95% CI 2-sided [9.97 to 20.68]

ADVERSE EVENTS:
Arm/Group | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 22/241
Other Adverse Events (participants affected / at risk) | 124/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=241)
Anaemia (Blood and lymphatic system disorders) | 1
Lung infection (Infections and infestations) | 1
Dystonia (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 1
Delusion of grandeur (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Hallucination, auditory (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 3
Schizoaffective disorder (Psychiatric disorders) | 4
Schizophrenia (Psychiatric disorders) | 4
Self injurious behaviour (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 2
Suicide attempt (Psychiatric disorders) | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal polyp (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=241)
Nausea (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 16
Decreased appetite (Metabolism and nutrition disorders) | 12
Akathisia (Nervous system disorders) | 15
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 24
Sedation (Nervous system disorders) | 17
Somnolence (Nervous system disorders) | 35
Anxiety (Psychiatric disorders) | 15
Insomnia (Psychiatric disorders) | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.